CLINICAL TRIAL: NCT06477497
Title: The Application of Comprehensive Prevention and Treatment Strategy of Placenta Accreta Spectrum Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Key Research and Development Program of China (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022YFC2704505
Record Dates: First submitted 2024-06-04; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Placenta Accreta Spectrum
Keywords: placenta accreta spectrum disorders
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Theoretical training, technical supporting and standardized referral process
- control group: usual care

SUMMARY:
Placenta accreta spectrum (PAS) disorders are pathological attachment of the placenta to myometrium, where trophoblastic cells invade the uterine placental interface. PAS can lead to severe postpartum hemorrhage or even maternal death. Prenatal diagnosis of PAS is essential for optimal obstetric management to improve the pregnancy outcomes. However, in some low resource regions in China, less than 20% PAS are detected before delivery.

To explore the feasibility and universality of the bundled prevention and treatment strategy for placenta accreta spectrum disorders in different levels of medical institutions, and to investigate its effectiveness in improving the specialized disease management capabilities of medical institutions at all levels. We will conduct a regional, cluster-randomized trial to assess a multicomponent PAS management strategy to improve the prepartum detection rate of PAS.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have regular prenatal examination at the research hospitals
* Pregnant women diagnosed with PAS before or after delivery

Exclusion Criteria:

* Pregnant women who have never been diagnosed with placental implantation disease throughout the pregnancy
* Pregnant women who were lost to follow-up during the study period

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with placenta accreta spectrum disorders
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
antepartum diagnosis rate of PAS | through study completion, an average of 1.5 year